CLINICAL TRIAL: NCT03322436
Title: A Non-interventional Patient Study to Demonstrate Medical Utility of the lncRNA to Predict HF in AMI Patients
Brief Title: HeartLinc, a Study With AMI Patients Undergoing PCI
Acronym: HeartLinc
Status: Completed | Type: Observational
Sponsor: Firalis SA (Industry)
Responsible Party: Sponsor
Other Study IDs: ST0083
Record Dates: First submitted 2017-10-24; First posted 2017-10-26 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: AMI Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and urine samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AMI patients treated by PCI: AMI patient treated by PCI at risk to develop Heart Failure
  Interventions: Diagnostic Test: HeartLinc kit

INTERVENTIONS:
Diagnostic Test: HeartLinc kit — Samples are collected and analyzed afterwards

SUMMARY:
HeartLinc is a non-interventional patient study to demonstrate medical utility of the lncRNA to predict HF in AMI patients. 300 patients are expected to be recruited.

DETAILED DESCRIPTION:
The recruiting phase of the study includes the recruitment of patients (36 months) and is followed by 12 month of monitoring for each patient. After deciding MI and PCI treatment by physical exam, ECG and other diagnostic methods, blood samples will be collected. After undergoing PCI, samples of the same patients will be collected during hospitalization days after PCI (D0-3) according to the patient study flowchart. After hospitalization, patients will be contacted by phone call or written questionary after 30 days (D30). After 6 and 12 months, patients are reinvited for a routine rehospitalisation to perform clinical exams and ECGs. Blood and urine samples will be collected after 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years
* Myocardial infarction in association with a recent acute coronary syndrome <24 hrs leading to a coronary angioplasty decision
* Myocardial infarction with ST-elevation (STEMI) or myocardial infarction following acute coronary syndrome without ST-segment shift with a significant elevation of non-ST troponin (NSTEMI)
* Participation in the Hearlink Cohort
* Collecting and signed informed consent for Heartlink study participation and consent to participate in the ancillary Heartlink 2 study

Exclusion Criteria:

* Sudden Cardiac arrest which resulted in resuscitation other than single, non-repeated electric shock,
* cardiogenic shock
* Severe extra-cardiac diseases involving the short-term life expectancy of patients (risk of death at one year
* Programmed major non-cardiac surgery
* Known Altered Left Ventricular function before Acute Coronary Syndrome inclusion
* History of left, right or global heart failure
* Significant heart failure at hospital admittance (KILLIP 2)
* Acute Coronary Syndrome know more than 24 hours
* History of Myocardial infarction
* Participation in any other in progress or stopped study for less than 3 months other than the Heartlink study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: AMI patients undergoing PCI
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2018-03-13 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
LV-EF < 40% | 12 months
  Proportion of patients with LV-EF < 40% at 12 months measured by echocardiography

SECONDARY OUTCOMES:
LVEDV | 12 months
  Left Ventricular End Diastolic Volume (LVEDV) at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Hüseyin FIRAT, MD, PhD,, Principal Investigator — Firalis SA
Locations (2):
- CHU de TOULOUSE, Toulouse, France
- SNUH, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No